CLINICAL TRIAL: NCT02518568
Title: Study of the Pharmacokinetics of Serum Iron After a Single Oral Administration of Ferrous Sulphate Supplement Synthetic Formula in Women With Iron Deficiency Anaemia.
Brief Title: Ferrous Sulphate Supplement (V0355) in Women With Iron Deficiency Anaemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V00355 CP 1 02; 2015-000544-42 (EudraCT Number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

ARMS (1):
- Drug (Experimental)
  Interventions: Drug: V0355

INTERVENTIONS:
Drug: V0355 — Oral administration (2 tablets)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of serum iron after a single oral administration of 160 mg (2 tablets of 80 mg) V0355 in women with iron deficiency anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years inclusive with iron deficiency anaemia
* haemoglobin level between 85 g/L and 105 g/L
* serum ferritin level < 15 µg/L
* D14 +/- 7 days of the menstruation cycle on the day of pharmacokinetic evaluation

Exclusion Criteria:

* Anaemia related to other causes than iron deficiency and particularly inflammatory anaemia, anaemia due to marrow failure, haemopathy, haemoglobinopathies (sickle cell disease, thalassemia), haemolytic anaemia, anaemia due to acute haemorrhage, or anaemia related to chronic renal failure,
* Haemochromatosis or iron overload of secondary origin (blood transfusion),
* Long term treatment known to modify iron absorption,
* Gastro duodenal ulcer,
* Inflammatory bowel disease or any digestive disease which could modify iron absorption,
* Serious or progressive disease (cardiac, pulmonary, hepatic, renal, haematological, malignancy, autoimmune disease, infectious disease or neuropsychiatric disorders),
* Surgery undergone within 1 month prior to selection visit or a surgery planned during the study realization.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma concentration (Cmax) | up to 24 hours after oral administration
Time to Maximum Concentration (Tmax) | up to 24 hours after oral administration
Area under the iron plasma concentration curve (AUC) | up to 24 hours after oral administration

SECONDARY OUTCOMES:
Tolerability of single administration | Up to 24 hours
  Tolerability by evaluating the number of subjects with emergent adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Sofia, Bulgaria
- Iași, Romania